CLINICAL TRIAL: NCT06171230
Title: Eye Movement Desensitization and Reprocessing (EMDR) as a Treatment for Chronic Painful Diabetic Peripheral Neuropathy
Acronym: EMDR4CPDN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dijklander Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC 090
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Neuropathic Pain; Diabetes Mellitus
MeSH Terms: conditions — Neuralgia; Diabetes Mellitus | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: A single-case experimental design, replicated nine times (N-of-1 study).
Masking Description: In psychological research, it is not feasible to employ a 'blind' approach for both participants and EMDR therapists regarding the intervention. An independent research assistant, not otherwise involved in the study, oversees the completion of daily measurements and questionnaires. This ensures that EMDR therapists remain blind to the obtained data. An exception to this is the utilization of the results from the LEC and PCL-5, which are employed for case conceptualization. There will be no randomization of baseline length or initiation of the intervention, as seen in multiple baseline designs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye Movement Desensitization and Reprocessing (Experimental): Participants will undergo six 90-minute EMDR sessions. The EMDR treatment concludes when the selected target images attain a Subjective Units of Disturbance (SUD) score of 0 or when three consecutive sessions show no further decrease in the SUD. Between the baseline phase (phase A) and the intervention phase (phase C), an attention control phase is introduced (phase B). This phase controls for the non-specific effects of the intervention, such as attention, treatment contact, and social support.
  Interventions: Other: Eye Movement Desensitization and Reprocessing; Other: Attention control phase

INTERVENTIONS:
Other: Eye Movement Desensitization and Reprocessing — Using the LEC and PCL-5, emotionally charged images are selected at the onset of the EMDR intervention. Initially, events meeting the criteria for PTSD (A-criterion worthy events) are processed. Subsequently, pain-related experiences, including any distressing images, are addressed. If the emotional charge of the events diminishes (SUD=0) before the completion of the six EMDR sessions, the participant is categorized as an 'early completer,' and the post-assessment is conducted immediately. The duration of each EMDR session is 90 minutes.
Other: Attention control phase — Prior to EMDR, there is a two-week attention control phase. During this phase, the participant is asked to daily record their activities, emotions, and thoughts when experiencing pain. This information is further explored and evaluated in two sessions lasting 45 minutes each, involving in-depth discussions with the participant.

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) therapy in reducing pain intensity in individuals with chronic painful diabetic neuropathy (PDN). The main questions it aims to answer are:

1. Does EMDR therapy significantly reduce pain intensity in individuals with chronic PDN?
2. What is the impact of EMDR therapy on secondary outcomes, specifically anxiety, sleep disturbances, and personalized pain-related limitations? Additionally, the study will explore the correlation between pain scores and symptoms of post-traumatic stress disorder (PTSD) in individuals with chronic PDN.

Participants will undergo EMDR therapy sessions, focusing on the processing of emotionally charged pain-related events and addressing the pain itself. Main tasks for participants include active engagement in EMDR therapy sessions. Treatment outcomes, including changes in pain intensity, anxiety levels, sleep quality, and personalized pain-related limitations, will be monitored throughout the study.

DETAILED DESCRIPTION:
The study adopts a single-case experimental design, replicated nine times (N-of-1 study).

Research on the effectiveness of EMDR therapy for neuropathic pain is limited to studies on phantom pain (and complex regional pain syndrome (CRPS). In the case of CRPS, two case reports are available, and for phantom pain, there is one RCT with 60 participants and three studies with 10 or fewer participants, without a control group. In the phantom pain studies, EMDR therapy focused on processing memories of events leading to the onset and exacerbation of pain (initial injury, amputation) and pain-related memories with current emotional charge. Sometimes, but not always, these events were life-threatening, as seen in PTSD (American Psychiatric Association Painful experiences, such as falling on the stump, or anticipated catastrophes (nightmares or disaster fantasies) with current emotional charge, were also processed. In the CRPS studies, EMDR therapy targeted traumatic events, including those from childhood, and pain-related events. In all studies, after the events were processed, pain itself was taken as the target for EMDR therapy. The studies demonstrate that after EMDR therapy, pain intensity decreases, as do comorbid symptoms.

Research on the effectiveness of EMDR therapy as a treatment for chronic PDN, to the best of our knowledge, has not been conducted. The aim of the presented study is to investigate the effect of EMDR therapy on chronic PDN.

ELIGIBILITY:
Inclusion criteria:

* Age: ≥ 18 years.
* Diagnosis of Diabetes Mellitus.
* Severity of pain in the past month, NRS-pain score ≥ 6.
* Ability to communicate in both written and spoken Dutch.
* Willingness to participate in the study (signed informed consent (IC)).

Exclusion criteria:

* Severe psychiatric disorders requiring immediate treatment.
* IQ < 80.
* Initiation of medication within 3 months before the start of the study (medication in use for more than 3 months can be maintained; discontinuation of medication during the study is possible but not desirable).
* Concurrent psychotherapeutic treatment targeting neuropathic pain during the study.
* Substance abuse and/or dependence, unless medically prescribed.
* Inability to complete the questionnaires.
* Co-morbid conditions affecting the lower extremities, such as peripheral arterial disease, severe rheumatoid arthritis, osteoarthritis. Other conditions causing pain in the feet and/or damage to the peripheral nervous system, for example, ulcers.
* Co-morbid chronic pain syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured with the Numeric Rating Scale (NRS) | Pain intensity is assessed once daily in the evening for a maximum of 154 days (throughout all phases of the study (phase A, phase B, phase C, post-assessment phase, and follow-up phase.)
  The NRS is an 11-point numeric scale form 0 (no pain ) to 10 (worst pain)

SECONDARY OUTCOMES:
Anxiety | The anxiety level is assessed once daily in the evening for maximum of 154 days (throughout all phases of the study (phase A, phase B, phase C, post-assessment phase, and follow-up phase.)
  Anxiety is scored on an 11-point scale from 0 (no anxiety) to 10 (most imaginable anxiety).
Quality of your sleep | Sleep problems are assessed once daily in the evening for a maximum of 154 days (throughout all phases of the study (phase A, phase B, phase C, post-assessment phase, and follow-up phase.)
  Sleep problems are scored on an 11-point scale from 0 (least possible sleep) to 10 (best possible sleep).
Pain Disability Index (PDI) Limitations in daily activities | The selected questions from the PDI are assessed once daily in the evening for a maximum of 154 days (throughout all phases of the study (phase A, phase B, phase C, post-assessment phase, and follow-up phase.)
  Two questions from the PDI, deemed most relevant by the participant, are chosen in collaboration with the participant. The limitations are scored on an 11-point scale from 0 (no limitations) to 10 (fully restricted).

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Zyto, Drs, Principal Investigator — Dijklander Ziekenhuis
Locations (1):
- Dijklander Ziekenhuis, Hoorn, Netherlands

IPD SHARING:
Plan to Share IPD: No